CLINICAL TRIAL: NCT05151159
Title: Prognostic Value of Protein IMP3 Expression in Cervical Cancer
Status: Completed | Type: Observational
Sponsor: University of Mostar (Other)
Responsible Party: Principal Investigator, Tanja Kresic, Mr.sc. Tanja Krešić, ob/gyn specialist, gyn oncology subspecialist, University of Mostar
Other Study IDs: IMP3, cervical cancer
Record Dates: First submitted 2021-11-23; First posted 2021-12-09 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Parts of cervix

GROUPS / COHORTS (4):
- FIGO group 1A1: 20 subjects with tumor invasion depth up to 1 mm
  Interventions: Other: immunohistochemical analysis with murine monoclonal antihuman antibodies IMP3
- FIGO group 1A2: 20 subjects with an invasion depth of 1 - 3 mm
  Interventions: Other: immunohistochemical analysis with murine monoclonal antihuman antibodies IMP3
- FIGO group 1B1: 20 subjects with invasion depth up to 2 cm
  Interventions: Other: immunohistochemical analysis with murine monoclonal antihuman antibodies IMP3
- FIGO group 1B2: 20 subjects with tumor invasion depth> 2 cm 20 subjects with tumor invasion depth> 2 cm
  Interventions: Other: immunohistochemical analysis with murine monoclonal antihuman antibodies IMP3

INTERVENTIONS:
Other: immunohistochemical analysis with murine monoclonal antihuman antibodies IMP3

SUMMARY:
The results of recent research on cervical cancer and its precancerous lesions have linked the expression of IMP3 protein to cervical dysplasia and the possibility of severe cervical dysplasia (CIN III) progressing to squamous cell carcinoma. A higher expression of IMP3 protein was found in the cytoplasms of severe cervical dysplasia (CIN III) cells and invasive tumor cells compared to CIN I and CIN II change cells. The sensitivity of IMP3 expression in tumor cells was 96%. In preparations that were IMP3 negative, no further monitoring and treatment revealed squamous cell carcinoma. Further analyzes indicated the possibility of determining IMP3 expression on first cervical biopsy specimens in patients with HSIL ( high grade squamous intraepithelial lesion) lesions as a biomarker to detect a subset of patients in whom lesion invasiveness can be expected.

DETAILED DESCRIPTION:
Molecular biomarkers could selectively identify patients with a more unfavorable clinical course. One of these biomarkers is IMP3 - insulin-like growth factor II mRNA binding protein.

The IGF group is a complex regulatory network at the cellular and substantial levels and plays a key physiological role in the development of the organism and the maintenance of normal cellular function during fetal and postnatal life. Overexpression of growth factors and their receptors is a common event during carcinogenesis. The IGF signaling system is under strict control of the normal physiological state and a deviation in this delicate balance can be a trigger for many molecular events leading to the development of malignancy. One member of the IGF system is the insulin-like growth factor II mRNA binding protein (IMP) which has been found to be an activator of IGF-II translation mRNA thus gaining a dominant role in controlling IGF-II-dependent cell proliferation.

The IMP protein family contains 3 proteins (IMP1, IMP2, IMP3). IMP3 is normally expressed in fetal tissues during embryogenesis. In adulthood, it appears as an oncoprotein that is expressed only in tumor tissues without the presence in the surrounding (adjacent) benign tissue. Previous in vitro studies have shown that IMP3 stimulates tumor cell proliferation by activating IGF II translation and adhesion and invasion via adhesion molecules and matrix metalloproteinases 1.

The results of recent research on cervical cancer and its precancerous lesions have linked the expression of IMP3 protein to cervical dysplasia and the possibility of severe cervical dysplasia (CIN III) progressing to squamous cell carcinoma. A higher expression of IMP3 protein was found in the cytoplasms of severe cervical dysplasia (CIN III) cells and invasive tumor cells compared to CIN I and CIN II change cells. The sensitivity of IMP3 expression in tumor cells was 96%. In preparations that were IMP3 negative, no further monitoring and treatment revealed squamous cell carcinoma. Further analyzes indicated the possibility of determining IMP3 expression on first cervical biopsy specimens in patients with HSIL lesions as a biomarker to detect a subset of patients in whom lesion invasiveness can be expected.

Based on previous studies, a monoclonal antibody specific for IMP3 has been developed and is successfully used in routine immunohistochemical methods that study the expression of IMP3 proteins in various malignancies. It has recently been found that the expression of IMP3 protein is associated with a more aggressive clinical course and a less favorable outcome in both gynecological and malignant diseases of other organ systems.

Research issues

Despite previous knowledge of prevention, detection and treatment, cervical cancer still causes great pain and mortality. The clinical course has so far been overlooked with regard to the clinical and pathological stage of the disease, and based on histological parameters and anatomical extent of the disease, a decision was made on further treatment and prognosis of the disease.

Previous research has only provided an introduction to the association of IMP3 protein expression with cervical cancer. An association was found between the increased expression of IMP3 protein in gynecological and other cancers in the body with a poorer disease outcome.

This study would look at the expression of IMP3 protein in cervical squamous cell carcinoma with the aim of detecting and linking the increased expression of IMP3 protein in patients who are expected to have an unfavorable clinical course and a poorer prognosis. Only patients in FIGO 1A1 and 1B1 disease stages will be observed, which has not been done in previous studies. In this way, patients who would be treated surgically would be singled out, and in whom a worse clinical outcome could be predicted and additional treatment could be planned individually.

Purpose of research

The study will determine the importance of immunohistochemical expression of IMP3 protein in cervical squamous cell carcinoma as a prognostic factor associated with higher tumor histological grade, higher FIGO stage, poorer course and disease outcome.

Reasearch hypothesis

Immunohistochemical expression of IMP3 protein in cervical squamous cell carcinoma was associated with poorer clinical course and disease outcome, shorter disease-free interval duration, and poorer 5-year survival outcomes.

Immunohistochemical determination of IMP3 protein expression in cervical cancer - as a new prognostic factor

The following will be excluded from the research:

* patients who have undergone pre-operative chemo and / or radiotherapy
* patients with associated gynecological or other malignancies
* patients with other histological types of tumors (adenocarcinoma, adenosquamous, neuroendocrine, etc.) The research will be performed on pathohistological preparations of surgical material of patients operated for cervical cancer in SKB Mostar in the above period.

The expression of IMP3 protein will be determined by immunohistochemical method and statistical analysis will be used to assess the association of expression with clinical and pathological disease progression and survival parameters.

Insight into medical documentation (patient medical histories and medical documentation of oncology patients from the Department of Oncology and Gynecology Clinic SKB Mostar) will provide clinical data on the age of patients, clinical stage of the disease determined by FIGO classification criteria, recurrence / length of period without signs of disease and clinical outcome.

Research methods:

Tumor samples for analysis will be obtained by 4μ sections of archived paraffin blocks.

Mouse monoclonal antihuman antibodies an IMP3 (DAKO) at a dilution of 1: 100 will be used for immunohistochemical analysis.

The immunohistochemical process will begin by dewaxing the tissue first in xylene and then rehydrating in alcohols of ever lower concentrations. Incubation in 0.1% H2O2 (30 minutes at room temperature) inactivated endogenous peroxidase. In order to detect antigenic sites, the sections will be boiled in citrate buffer, pH 9, in a microwave oven at 95 ° C for 10 minutes, then washed in phosphate buffered saline (PBS). After cooling to room temperature, the sections were incubated with primary antibodies for 60 minutes. After one hour of incubation with the primary antibody and washing in PBS, secondary detection with diaminobenzidine (DAB) will be used. An antibody-independent EnVision Detection Systems Peroxidase (DAB, Rabbit / Mouse K 5007) will be used for this purpose. After a 30-minute incubation and washing in PBS, the sections will be stained with diaminobenzidine (DAB) for 10 minutes at room temperature and washed in distilled water, and stained with hemalaun. The incisions will then be fitted into the fitting medium and covered with coverslips. Cells that reacted with the appropriate primary antibodies should have stained cytoplasms.

The results of immunohistochemical staining will be interpreted semiquantitatively. Samples with cytoplasmic staining in more than 10% of tumor cells will be considered as positive expression, and will be classified into 5 categories: 0 (1% -10% of stained cells), 1 (11% -25%), 2 (26% 50) %), 3 (51% -75%) and 4 (76% -100%). The intensity of IMP3 expression will be classified as negative, weak, moderate, or severe.

Sections intended for negative control by immunohistochemical staining of each antigen will be subjected, along with other sections, to the same procedure, except that they will not incubate with the primary antibody, but will be in PBS during that time. Control slides by the manufacturer will be used as a positive control.

The specimens will be examined with an Olympus BX40 light microscope (Olympus, Tokyo, Japan).

Total patient survival (OS) was defined as the time period between the date of surgery and the date of the last clinical control or death from cervical cancer.

Disease-free interval (DFS) is defined as the time interval between the date of surgery and the date of disease recurrence.

Statistical data processing:

The obtained research results will be stored in the MS Excel 2007 database, for all statistical analyzes the SPSS 17 statistical program will be used. Descriptive statistics methods will be used in data analysis. Nonparametric variables will be displayed as frequency and percentage. Depending on the data distribution, the parametric variables will be displayed as the arithmetic mean and standard deviation or as the median and interquartile range. The data distribution will be tested by the Kolmogorov-Smirnov test. A chi-square test and Fisher's exact test will be used to test for differences between groups for categorical variables where necessary. Student t-test and one-way analysis of variance (ANOVA) or Mann-Whitney U test and Kruskal-Wallis test as non-parametric alternatives in case the data distribution deviates from normal will be used to test the difference between parametric variables. Appropriate correlation and regression tests will be used to test the correlation between the examined variables. In the analysis of survival and disease recurrence, the Kaplan-Meier method and the Cox-Mantel log-rank test or the Mantel-Haenszel test will be used depending on the data obtained. The probability level of p <0.005 will be taken as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* operated women diagnosed with squamous cell carcinoma of the cervix at the figo stage 1a1, 1a2, 1b1 and 1b2

Exclusion Criteria:

* patients who underwent preoperative chemo and / or radiotherapy
* patients with associated gynecological or other malignant diseases
* patients with other histological types of tumors (adenocarcinoma, adenosquamous, neuroendocrine, etc.)

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Study Population: Operated women in University Clinic Mostar, who were diagnosed with squamous cell carcinoma cervicis in period of January 2003 to Decembar 2013.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
High expression of IMP3 protein in cervical squamous cell carcinoma is associated with a poorer disease outcome. | 10 Years ( 2003-2013)
  Investigators are about to examine the association between IMP3 protein expression and disease spread according to the FIGO classification (clinical-pathological grading of the disease)

CONTACTS AND LOCATIONS:
Overall Officials: Krešić Tanja, Mr.sc, Principal Investigator — University Mostar

IPD SHARING:
Plan to Share IPD: Yes
All of the individual Participant Data collected during the Trial.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning by three months and ending 5 Years following article publication.
Access Criteria: Investigators whose proposed use the Data has been approved by an Independent Review committe identified for this purpose.